CLINICAL TRIAL: NCT03829345
Title: A Translational Phase II Study of Single Agent Olaparib in the Treatment of Advanced Oesophagogastric Cancer
Brief Title: A Translational Study of Single Agent Olaparib in the Treatment of Advanced Oesophagogastric Cancer
Acronym: SOLAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR4825
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Oesophageal Cancer; Gastro-Oesophageal Junction Cancer; Gastric Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olaparaib (Experimental): Olaparib will be given 300mg bd for a 28 day cycle.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Patients will be administered olaparib orally twice daily (BD) at 300mg continuously for each 28 day cycle.

SUMMARY:
SOlar is a multi-centre phase II clinical trial of single agent olaparib in advanced oesophagogastric cancer.

DETAILED DESCRIPTION:
Gastric and oesophageal cancers are a significant health burden and are a leading cause of cancer related death. Despite improvements in survival over the last 4 decades overall the outcomes remain poor. In patients with advanced disease the outlook is particularly bleak with survival rates of less than one year with first line chemotherapy. New treatments are urgently needed to improve the poor survival rates in these cancers.

Olaparib is a PARP inhibitor which blocks poly(ADP-ribose) polymerase (PARP) 1, an enzyme which is involved in repair of damaged DNA. By inhibiting PARP1 olaparib prevents repair of damaged DNA. Cells with unrepaired DNA cannot survive and die.

This trial is designed to assess the efficacy and safety/tolerability of olaparib in patients with advanced oesophagogastric cancer. It will be conducted in two stages:

* The first stage will evaluate the efficacy of olaparib in 27 patients. If 4 or fewer patients have control of their disease at 8 weeks then the trial for the olaparib arm will stop and no further patients will be recruited to the study. If 5-13 patients have control of their disease at 8 weeks then the study will progress to stage 2. If 14 or more patients have disease control at 8 weeks then a larger study may be opened in an unselected population.
* The second stage will evaluate disease control in a further 27 patients. This is to allow identification of potential biomarkers of response.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced or metastatic oesophageal, gastro-oesophageal junction or gastric adenocarcinoma that has progressed during or within 6 months of first or subsequent line treatment
2. Patients with HER2-positive oesophageal, gastro-oesophageal, or gastric adenocarcinoma must have received previous treatment with trastuzumab
3. Male and female patients ≥18 years of age
4. Availability of tissue sample (resection or biopsy) confirming oesophageal, gastro-oesophageal junction, or gastric adenocarcinoma. If the patient does not have prior histological diagnosis, then the planned baseline fresh tumour biopsy may be used for both the purpose of confirming the histological diagnosis and subsequent biomarker analysis. All patients must be willing to have a fresh tumour biopsy to obtain tumour tissue for biomarker analysis at baseline and on progression
5. Disease amenable to safe biopsy
6. At least one lesion, not previously irradiated, that can be accurately measured as per RECIST criteria 1.1
7. Able to give informed consent
8. Adequate organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below: Hb 10.0 g/dL independent of blood transfusions for 28 days, Absolute neutrophil count (ANC) 1.5 x 109/L, Platelet count ≥ 100 x 109/L, INR < 1.5, Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN), AST/ ALT ≤ 2.5 x institutional ULN (unless liver metastases are present in which case it must be ≤ 5x ULN), Serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN) or a calculated creatinine clearance >51 mL/min for patients with creatinine levels above institutional normal. For GFR estimation, the Cockcroft and Gault equation should be used: GFR = CrCl (ml/min) = (140 - age [years]) × weight (kg) (xF)a /(serum creatinine [mg/dL]× 72)awhere F =0.85 for females and F=1 for males, Albumin >33 g/L
9. WHO ECOG performance status 0-1
10. Life expectancy of 16 weeks or more
11. Negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1) or postmenopausal status Postmenopausal status is defined as: Amenorrhoeic for 1 year or more following cessation of exogenous hormonal treatments, LH and FSH levels in the postmenopausal range for women under 50, Radiation induced oophorectomy with last menses >1 year ago, Chemotherapy-induced menopause with >1 year interval since last menses, Or surgical sterilisation (bilateral oophorectomy or hysterectomy)
12. Patient is willing and able to comply with the protocol for the duration of the study including having examinations, undergoing treatment, and attending scheduled visits (including follow up)
13. Patients of child bearing potential and their partners, who are sexually active, must agree to the use of TWO acceptable effective birth control methods in combination throughout their participation in the study and for at least 1 month after the last dose of study drug. For example, condom with spermicide and oral contraceptive/hormonal therapy or condom with spermicide and placement of an intra-uterine device.

Exclusion Criteria:

1. Any previous treatment with a PARP inhibitor, including olaparib
2. Any second primary cancer (except adequately treated non-melanoma skin cancer, curatively treated cervical carcinoma-in-situ and curatively treated other solid tumours with no evidence of disease for 5 years or more)
3. Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons) or investigational product within 4 weeks from the last dose prior to starting treatment (or a longer period depending on the defined characteristics of the agents used). A stable dose of bisphosphonates is permitted for bone metastases before and during the study as long as they were started at least 4 weeks prior to starting treatment
4. Clinically significant heart disease such as uncontrolled symptomatic arrhythmias, congestive heart failure, or myocardial infarction within the previous 3 months of screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
5. Interstitial pneumonia or symptomatic fibrosis of the lungs
6. Active brain or leptomeningeal metastases. A scan to confirm the absence of brain metastases is not required. Patients with known brain metastases are eligible if they have been treated and there is no evidence of progression for at least 4 weeks after treatment is complete and within 28 days prior to first dose of study drug administration. Patients can take a stable dose of corticosteroids before and during the study as long as these were started 4 or more weeks prior to treatment
7. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any previous major surgery
8. Pregnant and breastfeeding women
9. Patients considered a poor medical risk due to a serious uncontrolled medical disorder, non-malignant systemic disease or active uncontrolled infection. Examples include, but are not limited to, uncontrolled major seizure disorder, unstable spinal cord compression (untreated and unstable for at least 28 days prior to study entry), superior vena cava syndrome, extensive bilateral lung disease on HRCT scan or any psychiatric disorder that prohibits obtaining informed consent
10. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with study medication absorption
11. Persistent toxicities (of CTCAE grade 2 or above) with the exception of alopecia, caused by previous cancer therapy
12. Immunocompromised patients e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV)
13. Patients with known active hepatic disease (i.e. Hepatitis B or C)
14. Patients with intestinal obstruction or patients with CTCAE grade ≥ 3 upper GI bleeding within 4 weeks of study entry
15. Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
16. Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents
17. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
18. Previous enrolment in the present study
19. Resting ECG with QTc of over 500 msec on 2 or more time points within a 24 hour period or a family history of long QT syndrome.
20. Patients with myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML) or features suggestive of MDS/AML
21. Patients with known hypersensitivity to olaparib or any of the excipients of the products
22. Vaccinated with live, attenuated vaccines within 4 weeks of enrolment
23. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUBCT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-07-02 (Actual); Primary Completion 2021-02-14 (Estimated); Study Completion 2022-02-14 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate | 8 weeks from initiation of study drug
  The primary endpoint is disease control rate (DCR) defined as stable disease, partial response or complete response according to RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Doctor Starling, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Claire Saffery, Sutton, Surrey
  - Claire Saffery, Sutton

IPD SHARING:
Plan to Share IPD: Undecided